CLINICAL TRIAL: NCT04839419
Title: Prevalence of Obesity-hypoventilation Syndrome in Patients With Metabolic Syndrome.
Brief Title: Obesity-hypoventilation in Metabolic Syndrom Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SOS Oxygene Mediterranee (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-A02866-51
Record Dates: First submitted 2021-04-01; First posted 2021-04-09 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome; Obesity Hypoventilation Syndrome; Capnography
MeSH Terms: conditions — Metabolic Syndrome; Obesity Hypoventilation Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to determined the prevalence of obesity-hypoventilation syndrome in patients with metabolic syndrom.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, patient agreed to participate and undergo :

a functional respiratory exploration, an arterial blood gas analyze, and a polygraphy coupled with a capnography during the same night.

ELIGIBILITY:
Inclusion Criteria:

* BMI>30 kg/m2
* no treatment with CPAP nor NIV

Exclusion Criteria:

* obstructive respiratory disease
* non-treated cardiac dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be selected as part of their usual care, during a consultation for their respiratory and metabolic monitoring.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Capnia | Up to one mont after inclusion
  Arterial pression in CO2 and transcutaneous pression in CO2
Arterial pression in CO2 | At the inclusion
  PaCO2

SECONDARY OUTCOMES:
BMI | At the inclusion
  body mass index
Arterial pression in oxygen | At the inclusion
  PaO2
somnolence | At the inclusion
  EPWORTH questionnaire; Minimum = 0; Maximum = 24, Higher score means a worth outcome
Physical activity level | At the inclusion
  Ricci&Gagnon questionnaire, Minimum = 9; Maximum = 45, Higher score means a worth outcome
Arterial blood bicarbonates | At the inclusion
  HCO3-
Arterial blood gases | At the inclusion
  pH
Hemoglobin | At the inclusion
  Hb
obstructive sleep apnea items | Up to one mont after inclusion
  Apnea-hypopnea index
Night Oxygen saturation | Up to one mont after inclusion
  SpO2

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Despeaux, MD, Principal Investigator — Clinique du Chateau de Vernhes
Locations (1):
- Clinique du Château de Vernhes, Bondigoux, France